CLINICAL TRIAL: NCT05111912
Title: A Phase 2, Open-label, Randomised, Dose-Finding Study of XW003, Once-Weekly Human Glucagon-Like Peptide 1 Analogue, Compared With Once-Daily Liraglutide 3 mg in Adult Participants With Obesity
Brief Title: Effects of XW003 Versus Liraglutide on Body Weight of Adult Participants With Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sciwind Biosciences APAC CO Pty. Ltd. (Industry)
Collaborators: Hangzhou Sciwind Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCW0502-1121
Record Dates: First submitted 2021-10-17; First posted 2021-11-08 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort A (Experimental): Participants will follow a fixed up-titration scheme. For XW003 groups, the dose will be up-titrated to 1.2, 1.8, or 2.4 mg once weekly starting with 0.2 mg in dose increments of 0.2, 0.4, 0.6, or 0.8 mg. In order to mitigate the dose-related side effects, liraglutide is up-titrated over 4 weeks to the maintenance dose, 3.0 mg once daily.
  Interventions: Drug: XW003
- Cohort B (Experimental): Participants will follow a fixed up-titration scheme. For XW003 groups, the dose will be up-titrated to 1.2, 1.8, or 2.4 mg once weekly starting with 0.2 mg in dose increments of 0.2, 0.4, 0.6, or 0.8 mg. In order to mitigate the dose-related side effects, liraglutide is up-titrated over 4 weeks to the maintenance dose, 3.0 mg once daily.
  Interventions: Drug: XW003
- Cohort C (Experimental): Participants will follow a fixed up-titration scheme. For XW003 groups, the dose will be up-titrated to 1.2, 1.8, or 2.4 mg once weekly starting with 0.2 mg in dose increments of 0.2, 0.4, 0.6, or 0.8 mg. In order to mitigate the dose-related side effects, liraglutide is up-titrated over 4 weeks to the maintenance dose, 3.0 mg once daily.
  Interventions: Drug: XW003
- Cohort D (Active Comparator): Dose titration Saxenda (from 0.6 mg to 3.0 mg liraglutide once daily), should take place during the first 4 weeks after randomisation as described: Dose Escalation Schedule of Reference Product (Saxenda). All participants assigned to the open-labeled control group should aim to reach the final target dose of 3.0 mg liraglutide once daily.
  Interventions: Drug: Saxenda

INTERVENTIONS:
Drug: XW003 — XW003 (from 0.2 mg to 1.2 mg, 1.8 mg, and 2.4 mg once weekly), should take place during the first 14 weeks after randomization as described: Dose Escalation Schedule of Investigational Product (XW003). All eligible participants assigned to the XW003 study groups should aim to reach the respective final target dose of XW003 at 1.2 mg, 1.8 mg, or 2.4 mg once weekly.
  Other Names: GLP-1 analogue
  Arms: Cohort A; Cohort B; Cohort C
Drug: Saxenda — If a participant does not tolerate the recommended target dose of Saxenda group (e.g., 3.0 mg once daily), the participant may stay at the preceding highest tolerable dose (e.g., 2.4 mg once daily).
  Other Names: GLP-1 analogue
  Arms: Cohort D

SUMMARY:
XW003 is an acylated human glucagon-like peptide 1 (GLP-1) analogue and is being developed for type 2 diabetes mellitus (T2DM) and obesity management.

DETAILED DESCRIPTION:
The study treatment period for 4 groups in the study will be divided into the four Titration Treatment periods and one Core Treatment period. The overall duration of the study treatment for each group will be 26 weeks. The duration of Titration Treatment will be up to 14 weeks for the three groups of XW003 treatment but 4 weeks for Saxenda group.

Approximately 250 participants who are adults with obesity, in the absence of type 2 or any other type of diabetes, are planned to be screened. Based on a 20% screening failure rate, a total of 200 participants are expected to be enrolled for the four groups.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this study, a participant has to meet all of the following inclusion criteria:

1. Male or female, aged 18 to 70 years (inclusive at the time of informed consent);
2. Participants must have a BMI ≥ 30.0 kg/m2 and ≤40.0 kg/m2 at Screening;
3. Participants must have a stable body weight for at least 3 months prior to Screening (<5% change, self-reported);
4. Participants must have glycated haemoglobin (HbA1c) level <6.5% at Screening;
5. Women of childbearing potential (WOCBP) must be non-pregnant and must use an acceptable, highly effective contraception from Screening until the study completion, including the follow-up period.
6. Participants must have the ability and willingness to attend the necessary visits to the clinical research unit (CRU);
7. Participants must be willing and able to provide written informed consent after the nature of the study has been explained and prior to the commencement of any study procedures.

Exclusion Criteria:

A participant who meets any of the following exclusion criteria must be excluded from the study:

1. Diagnosis of type 2 (HbA1c ≥6.5%) or other types of diabetes mellitus;
2. Obesity induced by endocrine disorders (e.g., Cushing syndrome);
3. Calcitonin ≥50 ng/L (pg/mL) at Screening;
4. History of severe allergic or hypersensitivity to any of the investigational products or its excipients or to drugs of similar chemical classes;
5. History of cerebral stroke (including but not limited to cerebral infarction/haemorrhage) within 6 months prior to Screening;
6. History of acute coronary syndrome (angina pectoris and/or myocardial infarction) and any other major cardiac conditions (including but not limited to myocarditis, cardiac insufficiency/failure, and any clinically significant arrythmia[s]) within 6 months prior to Screening;
7. Impaired liver function defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >5 times upper limit of normal (ULN) at Screening;

Main Inclusion Criteria:

To be eligible for this study, a participant has to meet all of the following inclusion criteria:

1. Male or female, aged 18 to 70 years (inclusive at the time of informed consent);
2. Participants must have a BMI ≥ 30.0 kg/m2 and ≤40.0 kg/m2 at Screening;
3. Participants must have stable body weight for at least 3 months prior to Screening (<5% change, self-reported);
4. Participants must have glycated hemoglobin (HbA1c) level <6.5% at Screening;
5. Women of childbearing potential (WOCBP) must be non-pregnant and must use an acceptable, highly effective contraception from Screening until the study completion, including the follow-up period.
6. Participants must have the ability and willingness to attend the necessary visits to the clinical research unit (CRU);
7. Participants must be willing and able to provide written informed consent after the nature of the study has been explained and prior to the commencement of any study procedures.

Main Exclusion Criteria:

A participant who meets any of the following exclusion criteria must be excluded from the study:

1. Diagnosis of type 2 (HbA1c ≥6.5%) or other types of diabetes mellitus;
2. Obesity induced by endocrine disorders (e.g., Cushing syndrome);
3. Calcitonin ≥50 ng/L (pg/mL) at Screening;
4. History of severe allergic or hypersensitivity to any of the investigational products or its excipients or to drugs of similar chemical classes;
5. History of cerebral stroke (including but not limited to cerebral infarction/haemorrhage) within 6 months prior to Screening;
6. History of acute coronary syndrome (angina pectoris and/or myocardial infarction) and any other major cardiac conditions (including but not limited to myocarditis, cardiac insufficiency/failure, and any clinically significant arrythmia[s]) within 6 months prior to Screening;
7. Impaired liver function defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >5 times upper limit of normal (ULN) at Screening;
8. Estimated glomerular filtration rate (eGFR), calculated using the modified diet in renal disease (MDRD) formula < 60 mL/min/1.73m2;
9. History of acute or chronic pancreatitis or defined as amylase >ULN at Screening;
10. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2 (MEN2);
11. Positive infection with human immunodeficient virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV);
12. History of primary or recurrent malignancy, except for non-melanoma skin cancer excised more than 2 years prior to Screening;
13. History of clinically significant endocrine condition(s);
14. History of major depressive disorder within 2 years before randomisation;
15. History of surgical treatment for obesity;
16. Having been exposed to any GLP-1 analogues within 6 months before Screening;
17. Treatment with orlistat, zonisamide, topiramate, phentermine, lorcaserin, bupropion and naltrexone alone or in combination or any other medications that could promote weight loss within 90 days prior to Screening;
18. Use of any other investigational products or medical devices within 3 months prior to Screening;
19. Participation in any medical (e.g., assisted by a clinical dietician or nutritionist) or non-medical (e.g., by a gym coach) diet and/or exercise program within 3 months prior to Screening and for the duration of the study (including the follow-up period);
20. Known or suspected abuse of alcohol or recreational drugs;
21. Being pregnant or lactating at Screening or planning to become pregnant (self or female partner) at any time during the study and for at least 3 months after the last dose of study drug;
22. Presence of any underlying physical and/or psychological medical condition that, in the opinion of the investigator, would make it unlikely that the participant will comply with the protocol or complete the study per protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Percentage change in participants body weight (%) from the Baseline | Week 26
  Analysis of covariance (ANCOVA), with treatment, baseline body weight, and stratification factor as covariate, will be used to determine the difference between one of the XW003 groups and Saxenda group.

SECONDARY OUTCOMES:
Proportions of participants with body weight loss ≥5%, ≥10% and ≥15% of the Baseline | Week 26
  It is anticipated that XW003 can achieve considerable body weight loss and improve obesity-related markers in participants with obesity.
Absolute change in body weight (kg) of participants | Week 26
  Body weight should be measured at all site visits without shoes, on an empty bladder and only wearing light clothing.
Changes in waist circumference and hip circumference (cm) in participants | Week 26
  The waist circumference will be measured at the specified visits and is defined as the abdominal circumference located the midpoint between the lower rib margin and the iliac crest. The hip circumference is defined as the widest circumference around the buttocks.
Change in BMI in participants | Week 26
  Calculated by dividing the participant's body weight in kilograms by the participant's height in meters squared (kg/m2)
Change in fasting plasma glucose (FPG) | Week 26
  Calculated based on XW003 measured in blood.
Change in fasting serum insulin | Week 26
  Calculated based on XW003 measured in blood.
Change in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | Week 26
  Change in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR)
Changes in fasting lipids (triglyceride, low-density lipoprotein [LDL], and high-density lipoprotein [HDL]) | Week 26
  Lipids: triglyceride, low-density lipoprotein [LDL], and high-density lipoprotein [HDL].
Number and severity of treatment-emergent adverse events (TEAEs) | Week 26
  The most common treatment-emergent adverse events (TEAEs) were nausea, dyspepsia, constipation, vomiting, and loss of appetite, all of which deemed possibly related to XW003 injection and only occurred in the highest dose groups (0.6 mg and 1.0 mg). The severity of these TEAEs was mild or moderate.
Number and severity of new and ongoing gastrointestinal (GI) disorder (nausea, vomiting, diarrhea, and constipation) events by week | Week 26
  Analysis of the safety profile and tolerability of XW003 showed that the most common adverse events (AEs) of XW003 was gastrointestinal (GI) disorder, including nausea, bloating, loss of appetite, and weight loss.
Vital signs - participants' blood pressure change | Week 26
  After resting in a supine position for at least 5 minutes, the participant's systolic and diastolic blood pressure change.
Vital signs - participants' pulse rate change | Week 26
  After resting in a supine position for at least 5 minutes, the participant's pulse rate, and body temperature.
Vital signs - participants' ody temperature change | Week 26
  After resting in a supine position for at least 5 minutes, the participant's body temperature change.
Electrocardiograms (ECGs) | Week 26
  There was no XW003 injection related clinically significant effect 12-lead electrocardiography (ECG).
Haematology, biochemistry, coagulation, and calcitonin | Week 26
  Parameters to be tested are:
  * Haemoglobin (HGB)
  * Haematocrit (HCT)
  * Erythrocytes (RBC)
  * Platelets (PLAT)
  * Leucocytes (WBC) with differential
  * Urea
  * Creatinine (CREAT)
  * Total Bilirubin (BILI) and direct bilirubin (BILIDIR)
  * Urate
  * Albumin (ALB)
  * Alkaline phosphatase (ALP)
  * Creatine kinase (CK)
  * Alanine aminotransferase (ALT)
  * Aspartate aminotransferase (AST)
  * Gamma-glutamyl transferase (GGT)
  * Sodium (NA)
  * Potassium (K)
  * Calcium (CA)
  * Chloride (CL)
  * Phosphate (PHOS)
  * Bicarbonate (BICARB)
  * Amylase
  * Lipase
  * International Normalised Ratio (INR)
  * Activated partial thromboplastin time (APTT)
Injection site reactions (ISRs) | Week 26
  There were no hypoglycaemic episodes reported during the trial. Injection site reaction (ISRs) were reported in 1 participant in Cohort A2 (0.2/0.25 mg) and 2 participants in Cohort A6 (0.6 mg).
  The ISRs were mild in severity and recovered within 3 hours of dosing.
Physical examinations | Week 26
  It should include general appearance, thyroid gland, respiratory system, cardiovascular system, gastrointestinal system including mouth, musculoskeletal system, central and peripheral nervous system, skin, lymph node palpation, and head, ears, eyes, nose, throat and neck.
36-Item Short Form Survey (SF-36) | Week 26
  Physical and mental component summary scores and scores on the individual sub-domains, i.e., physical functioning, role functioning, bodily pain, general health, vitality, social functioning, role emotional and mental health

OTHER OUTCOMES:
Plasma concentrations of XW003 on treatment | Week 26
  Calculated based on XW003 measured in blood.
Anti-XW003 antibodies on treatment | Week 26
  Calculated based on XW003 measured in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Sheetal Bull, Principal Investigator — Paratus Clinical
Locations (1):
- Paratus Clinical Research Brisbane, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No